CLINICAL TRIAL: NCT05067140
Title: A Phase 1/2 Open-Label, Dose-Escalation and Cohort Expansion Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ARV-766 Monotherapy and in Combination With Abiraterone in Patients With Metastatic Prostate Cancer
Brief Title: A Study of ARV-766 Given by Mouth in Men With Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CJSB462A12101; ARV-766-mCRPC-101 (Other: Arvinas Inc.)
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer Metastatic
Keywords: Metastatic Prostate Cancer; Castrate-Resistant; Prostate Cancer; mCRPC adenocarcinoma of prostate; Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms; Castrate-Sensitive; mCSPC adenocarcinoma of prostate
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Urogenital Neoplasms | interventions — Adrenal Cortex Hormones; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARV-766 (Experimental): Oral tablets, once daily in 28 day cycles
  Interventions: Drug: ARV-766 Part A&B
- ARV-766 + Abiraterone (Experimental): Oral tablets, once daily in 28 day cycles
  Interventions: Drug: ARV-766 + Abiraterone Part C&D

INTERVENTIONS:
Drug: ARV-766 Part A&B — Part A: Daily oral dosages are determined by cohort review committee after initial starting dose cohort and each subsequent cohort completes 28 days of treatment.
  Part B: Oral tablet(s) once daily in 28 day cycles.
  Arms: ARV-766
Drug: ARV-766 + Abiraterone Part C&D — Part C: Daily oral combination dosages are determined by cohort review committee after initial starting dose cohort and each subsequent cohort completes 28 days of treatment.
  Part D: Combination administered once daily in 28 day cycles.
  Parts C&D: Participants will also receive concomitant corticosteroid and ADT therapy of investigator choice/patient preference
  Other Names: Corticosteroid and ADT
  Arms: ARV-766 + Abiraterone

SUMMARY:
A Phase 1/2 study to evaluate the safety and efficacy of ARV-766 given by mouth alone or in combination with abiraterone in men with metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

Part A,B,C and D:

* Histological, pathological, or cytological confirmed diagnosis of adenocarcinoma of the prostate.
* Ongoing androgen deprivation therapy (ADT) with a gonadotropin releasing hormone analog or inhibitor, or orchiectomy (surgical or medical castration).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Part A:

* Progression on at least 2 prior approved systemic therapies for metastatic prostate cancer (at least one must be a second-generation androgen inhibitor, e.g., abiraterone, enzalutamide, darolutamide, apalutamide).
* Progressive mCRPC

Part B:

* Participants must have received at least one but no more than three prior second generation anti-androgen agents (e.g., enzalutamide or abiraterone).
* Participants must have received no more than two prior chemotherapy regimens.
* Progressive mCRPC

Part C & D:

• Metastatic castration resistant or sensitive prostate cancer with radiographic evidence of metastatic disease

Exclusion Criteria:

Part A and B:

* Known symptomatic brain metastases requiring steroids (above physiologic replacement doses).
* Active inflammatory gastrointestinal disease, chronic diarrhea, known diverticular disease, or previous gastric resection or lap band surgery.
* Radiation therapy within 4 weeks of first dose of study drug or prior irradiation to >25% of the bone marrow.
* Receipt of an investigational drug(s) within 4 weeks prior to anticipated first dose
* Systemic anti-cancer therapy within 2 weeks of first dose of study drug (except agents to maintain castrate status). For bicalutamide, mitomycin C, or nitrosoureas the exclusion period must be 6 weeks and for abiraterone 4 weeks.

Part C and D

• Prior treatment with a second generation NHA

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 152 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2027-05-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Part A: Incidence of Dose Limiting Toxicities of ARV-766 | 28 Days
  First Cycle Dose limiting toxicities characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), timing, seriousness, and relationship to study drug
Part A: Number of Patients with Adverse Events as a measure of safety and tolerability of ARV-766 | 28 Days
  Adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), timing, seriousness, and relationship to study drug.
Part A: Incidence of laboratory abnormalities as a measure of safety and tolerability of ARV-766 | 28 Days
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), and timing.
Part B: To evaluate the clinical anti-tumor activity of ARV-766 in patients with mCRPC | 12 Weeks
  Evaluate PSA in patients with mCRPC in both dose groups
Part C: Incidence of Dose Limiting Toxicities of ARV-766 / abiraterone combination | 28 Days
  First Cycle Dose limiting toxicities characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), timing, seriousness, and relationship to study drug
Part C: Incidence of laboratory abnormalities as a measure of safety and tolerability of ARV-766 / abiraterone combination | 28 Days
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), and timing.
Part C: Number of Patients with Adverse Events as a measure of safety and tolerability of ARV-766 / abiraterone combination | 28 Days
  Adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE v 5.0), timing, seriousness, and relationship to study drug.
Part D: To evaluate the clinical anti-tumor activity of ARV-766 / abiraterone combination in patients with NHA-naïve mPC | 12 Weeks
  Evaluate PSA in patients with NHA-naïve mPC

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (23):
  - Clinical Trial Site, Duarte, California
  - Clinical Trial Site, Fresno, California
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Orange, California
  - Clinical Trial Site, Santa Monica, California
  - Clinical Trial Site, New Haven, Connecticut
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Lake Mary, Florida
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, New Orleans, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Buffalo, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Myrtle Beach, South Carolina
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Charlottesville, Virginia
  - Clinical Trial Site, Fairfax, Virginia
  - Clinical Trial Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No